CLINICAL TRIAL: NCT07168005
Title: Does an Informative Video Reduce Anxiety and Pain Before LMWH Treatment Postpartum? - A Randomized Controlled Trial
Brief Title: Informative Video Before LMWH Postpartum - Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0121-25-WOMC
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Venous Thromboembolism (VTE); Postpartum Care; Anxiety
Keywords: Postpartum; Venous Thromboembolism; VTE; LMWH; Low Molecular Weight Heparin; Clexane; Anxiety; Pain; Patient Education; Informative Video; State-Trait Anxiety Inventory; STAI; Postpartum Care; Women's Health; Obstetrics; Adherence
MeSH Terms: conditions — Venous Thromboembolism; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either the intervention group (standard explanation plus a short informative video) or the control group (standard explanation only). Both groups will receive their assigned explanation prior to the first postpartum LMWH (Clexane) injection. Outcomes will be assessed immediately following the intervention.
Masking Description: This is an open-label study. Neither participants nor healthcare providers are blinded to group allocation, as the nature of the intervention (informative video) makes blinding infeasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video (Experimental): Participants in this group will view a short (up to 5 minutes) informative video. The video explains the rationale, procedure, and safety of LMWH to reduce anxiety and increase patient understanding prior to the first injection.
  Interventions: Behavioral: Informative Video on LMWH
- Control Group (Active Comparator): Participants in this group will receive only a verbal explanation regarding postpartum LMWH (Clexane) administration, without any additional video intervention. This represents the current standard of care
  Interventions: Behavioral: Standard Verbal Explanation

INTERVENTIONS:
Behavioral: Informative Video on LMWH — A short (up to 5 minutes) informative video presented to postpartum women prior to their first LMWH (Clexane) injection. The video explains the rationale, process, and safety of LMWH use for thrombopr
  Arms: Video
Behavioral: Standard Verbal Explanation — Participants receive the routine verbal explanation regarding postpartum LMWH (Clexane) administration, covering its purpose and method of injection
  Arms: Control Group

SUMMARY:
This single-center randomized controlled trial evaluates whether a short informative video can reduce anxiety and pain before the first postpartum administration of low molecular weight heparin (LMWH, Clexane). Eligible women will be randomized to receive either standard explanation alone or standard explanation plus a short educational video. The primary outcome is anxiety level assessed via the State-Trait Anxiety Inventory (STAI). Secondary outcomes include pain, satisfaction, and treatment adherence.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a leading cause of maternal morbidity and mortality, with the postpartum period carrying a particularly elevated risk. As part of standard care, low molecular weight heparin (LMWH), typically Clexane, is frequently prescribed postpartum for thromboprophylaxis. However, the initiation of LMWH injections during the early postpartum period may provoke anxiety and discomfort due to heightened pain sensitivity, unfamiliarity with the treatment, and emotional vulnerability.

While informative videos have been shown to reduce patient anxiety and increase procedural satisfaction in various medical contexts, no studies have explored their use in the postpartum setting specifically for LMWH initiation. This study aims to determine whether a brief educational video shown to women prior to their first LMWH injection postpartum can reduce anxiety and pain, improve satisfaction, and potentially enhance adherence to treatment.

This is a prospective, single-center randomized controlled trial conducted at Edith Wolfson Medical Center. Women aged 18-45 who delivered at the hospital and are indicated for LMWH will be recruited and randomized in a 1:1 ratio into two groups. The control group will receive the standard verbal explanation from nursing staff regarding LMWH administration. The intervention group will receive the same standard explanation, followed by a short (up to 5 minutes) educational video explaining the rationale, process, and safety of LMWH therapy in the postpartum period.

The primary outcome is the anxiety level measured using the State-Trait Anxiety Inventory (STAI) after receiving the explanation or video and before the first LMWH injection. Secondary outcomes include the change in anxiety (ΔSTAI) before and after the intervention, pain and discomfort measured by an 11-point Visual Analog Scale (VAS), satisfaction with the explanation process, and adherence to LMWH treatment post-discharge as assessed via telephone follow-up.

The study will enroll 160 participants to account for an estimated 30% dropout rate, based on a calculated sample size of 126 participants needed to detect a clinically significant 5-point difference in STAI scores (power 80%, α = 0.05). Randomization will be performed using sealed envelopes. Blinding is not applicable. Data will be collected via structured questionnaires administered before and after the intervention, with follow-up data obtained via phone contact for those discharged with ongoing LMWH therapy.

Ethical approval will be obtained from the institutional review board prior to recruitment. Participation is voluntary, and informed consent will be obtained from all participants. All data will be anonymized and stored securely on password-protected hospital servers. No biological samples will be collected.

This study seeks to provide evidence on the role of simple digital educational tools in improving the postpartum care experience and reducing patient distress during routine pharmacologic interventions.

ELIGIBILITY:
Inclusion Criteria:

Women 18-45 years, postpartum, indicated for LMWH, Hebrew-literate, gave consent

Exclusion Criteria:

Use of LMWH pre-delivery, IUFD, pregnancy termination, language/cognitive barrier

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 160 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Post-intervention Anxiety Level (STAI Score) | Immediately after intervention and before first LMWH injection
  Anxiety will be measured using the State-Trait Anxiety Inventory (STAI) after participants receive either the standard explanation alone or view informative video, and before their first LMWH (Clexane) injection.

SECONDARY OUTCOMES:
Change in Anxiety Level (Δ STAI Score) | From baseline (before intervention) to immediately after intervention (within 1 hour postpartum)
  The difference in State-Trait Anxiety Inventory (STAI) score before and after the intervention (video or standard explanation) will be calculated to assess the change in anxiety levels.
Pain and Discomfort During Injection (VAS Score) | Immediately after the first LMWH injection
  Pain and discomfort will be assessed immediately after the first LMWH (Clexane) injection using an 11-point Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst possible pain).
Satisfaction With Explanation Process (VAS Score) | Immediately after the intervention and first injection
  Participants will rate their satisfaction with the explanation process (standard verbal vs. video-enhanced) using an 11-point Visual Analog Scale (VAS), ranging from 0 (not satisfied at all) to 10 (very satisfied).
Adherence to LMWH at Home | Up to 6 weeks post-discharge
  Among participants discharged with instructions for continued LMWH use, adherence will be assessed via structured telephone follow-up (self-reported number of injections taken vs. prescribed).

CONTACTS AND LOCATIONS:
Overall Officials: Matan Friedman, MD, Principal Investigator — Wolfson Medical Center; Amihai Rottenstreich, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) to be shared will include baseline demographics, STAI scores (pre- and post-intervention), Visual Analog Scale (VAS) scores for pain and satisfaction, and adherence data collected during follow-up. No personally identifying information will be included.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start Date: 6 months after publication of the primary results. End Date: 5 years after publication.
Access Criteria: De-identified individual participant data (IPD) and supporting documents (study protocol, statistical analysis plan, informed consent form) will be made available to qualified researchers affiliated with academic or healthcare institutions. Access will be granted upon reasonable request, subject to approval by the principal investigator and the Edith Wolfson Medical Center institutional review board. Approved data will be shared through a secure institutional file transfer system.

REFERENCES:
- [Background] MacLean S, Mulla S, Akl EA, Jankowski M, Vandvik PO, Ebrahim S, McLeod S, Bhatnagar N, Guyatt GH. Patient values and preferences in decision making for antithrombotic therapy: a systematic review: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e1S-e23S. doi: 10.1378/chest.11-2290. PMID 22315262
- [Background] Wong AKC, Chu RYK, Nan Y, Cheng H, Tong D, Leung M, Lam H, Chiu SH, Cheung HW, Chan MC, Chau MY, Lee T, Leung YW, Mow HC, Wan S, Wong LY, Montarye J. Injection Techniques to Reduce Adverse Effects of Subcutaneous Low-Molecular-Weight Heparin Among Patients With Cardiovascular Diseases: A Scoping Review. J Adv Nurs. 2025 Nov;81(11):7361-7373. doi: 10.1111/jan.16475. Epub 2024 Sep 25. PMID 39323021
- [Background] Middeldorp S, Ganzevoort W. How I treat venous thromboembolism in pregnancy. Blood. 2020 Nov 5;136(19):2133-2142. doi: 10.1182/blood.2019000963. PMID 32797192
- [Background] James AH. Prevention and management of venous thromboembolism in pregnancy. Am J Med. 2007 Oct;120(10 Suppl 2):S26-34. doi: 10.1016/j.amjmed.2007.08.011. PMID 17916457
- [Background] Bates SM, Rajasekhar A, Middeldorp S, McLintock C, Rodger MA, James AH, Vazquez SR, Greer IA, Riva JJ, Bhatt M, Schwab N, Barrett D, LaHaye A, Rochwerg B. American Society of Hematology 2018 guidelines for management of venous thromboembolism: venous thromboembolism in the context of pregnancy. Blood Adv. 2018 Nov 27;2(22):3317-3359. doi: 10.1182/bloodadvances.2018024802. PMID 30482767